CLINICAL TRIAL: NCT06910553
Title: CorEvitas Inflammatory Bowel Disease Pregnancy Registry (IBD-PR)
Brief Title: IBD Pregnancy Registry
Acronym: IBD-PR
Status: Recruiting | Type: Observational
Sponsor: CorEvitas (Network)
Responsible Party: Sponsor
Other Study IDs: IBDPR-310
Record Dates: First submitted 2025-03-06; First posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Inflammatory Bowel Disease (IBD)
Keywords: Pregnant; IBD; Registry; UC; Inflammatory Bowel Disease; Ulcerative Colitis
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (2):
- IBD pharmacotherapy exposed: Individuals with a diagnosis of IBD who are exposed to an approved IBD pharmacotherapy at any time during pregnancy
  Interventions: Drug: Exposed to IBD pharmacotherapy during pregnancy
- IBD pharmacotherapy unexposed: Individuals with a diagnosis of IBD who are not exposed to IBD pharmacotherapy during pregnancy
  Interventions: Other: Non-exposed group

INTERVENTIONS:
Other: Non-exposed group — Pregnant individuals with IBD who are not exposed to an IBD pharmacotherapy during pregnancy
  Groups: IBD pharmacotherapy unexposed
Drug: Exposed to IBD pharmacotherapy during pregnancy — Pregnant individuals with IBD who are exposed to an IBD pharmacotherapy during pregnancy
  Groups: IBD pharmacotherapy exposed

SUMMARY:
Data collected through the registry may be used to address a range of research questions and objectives, including but not limited to the following:

Research question: Is there an increased risk of adverse maternal, fetal, or infant outcomes among individuals who are exposed to Inflammatory Bowel Disease (IBD) treatments during pregnancy?

The primary objective of the registry is to estimate the prevalence of major congenital malformations among pregnant individuals with IBD who are exposed to an IBD pharmacotherapy during pregnancy.

The secondary objectives of the registry are:

To estimate the prevalence of other maternal, fetal, and infant outcomes among pregnant individuals with IBD who are exposed to IBD pharmacotherapies during pregnancy.

To contextualize the prevalence of outcomes among pregnant individuals who are exposed to IBD pharmacotherapies during pregnancy and estimate the prevalence of all outcomes of interest among pregnant individuals with IBD who are not exposed to any IBD pharmacotherapies or an IBD pharmacotherapy of interest during pregnancy.

If sample size permits, to estimate the risk ratio for each outcome, comparing the outcomes of pregnant individuals with IBD who are exposed to IBD pharmacotherapy with those who are not exposed to any IBD pharmacotherapies or an IBD pharmacotherapy of interest during pregnancy.

Data collection may be used to determine pharmacotherapy-specific use with or without unexposed cohorts on an as-needed basis, as sample size allows.

DETAILED DESCRIPTION:
Rationale and Background:

Inflammatory bowel disease (IBD) is a group of chronic inflammatory conditions that affect the gastrointestinal tract and can be divided into two main types: Crohn's disease (CD) and ulcerative colitis (UC). Half of the people diagnosed with IBD received their diagnosis before the age of 35 years, which coincides with the peak reproductive years for women. Studies have shown that IBD is associated with increased risk of adverse pregnancy and fetal outcomes, including preterm birth, stillbirth, and low birth weight. The CorEvitas IBD Pregnancy Registry (IBD-PR) aims to collect real-world evidence on the safety of IBD pharmacotherapies during pregnancy and the first year of infant life and provide valuable insights into the risks and safety profiles of IBD medications, enabling healthcare professionals to make more informed decisions when managing IBD in pregnant individuals.

Research Question and Objectives: Data collected through the registry may be used to address a range of research questions and objectives, including but not limited to the following:

The research question is: Is there an increased risk of adverse maternal, fetal, or infant outcomes among individuals who are exposed to IBD pharmacotherapies during pregnancy?

The primary objective of the registry is to estimate the prevalence of major congenital malformations (MCM) among pregnant individuals with IBD who are exposed to an IBD pharmacotherapy during pregnancy.

The secondary objectives of the registry are:

To estimate the prevalence of other maternal, fetal, and infant outcomes among pregnant individuals with IBD who are exposed to an IBD pharmacotherapy during pregnancy

To contextualize the prevalence of outcomes among pregnant individuals who are exposed to IBD pharmacotherapies during pregnancy and estimate the prevalence of all outcomes of interest among pregnant individuals with IBD who are not exposed to an IBD pharmacotherapy during pregnancy

If sample size permits, to estimate the risk ratio for each outcome, comparing the outcomes of pregnant individuals with IBD who are exposed to an IBD pharmacotherapy with outcomes of those who are not exposed to an IBD pharmacotherapy

Data collection may be used to determine pharmacotherapy-specific use with or without unexposed cohorts on an as-needed basis, as sample size allows.

Study Design: This prospective, observational cohort study is designed to estimate the prevalence of maternal, fetal, and infant outcomes among individuals with IBD who are exposed to an IBD pharmacotherapy during pregnancy. For this registry, the index date will be the date of first exposure to the IBD pharmacotherapy for the exposed cohort and the date of enrollment for the unexposed cohort. The risks of pregnancy-related outcomes, maternal outcomes, and neonatal/infant outcomes will be estimated for participants with IBD exposed and unexposed to any IBD pharmacotherapies or an IBD pharmacotherapy of interest during pregnancy.

Population: The registry population will include two cohorts of pregnant individuals: one cohort of individuals with a diagnosis of IBD who are exposed to an IBD pharmacotherapy during pregnancy and one cohort of individuals with a diagnosis of IBD who are not exposed to IBD pharmacotherapies during pregnancy.

Variables: Individuals will be considered exposed during pregnancy if at least one dose of an IBD treatment is taken during pregnancy or up to at least five times the product's half-life before conception. The primary outcome of interest is MCMs. The maternal and pregnancy secondary outcomes include minor congenital malformations, preeclampsia, eclampsia, spontaneous abortion, stillbirth, pregnancy termination, preterm birth, small for gestational age, gestational diabetes, pregnancy-induced hypertension, and placental abruption. The infant secondary outcomes during the first year of life include postnatal growth deficiency, infant developmental delay, infant hospitalization, infant infections (both serious and nonserious), and infant death. Covariates will include demographics, risk factors for the outcomes, comorbidities, concomitant medications, and predictors of treatment with an approved IBD pharmacotherapy.

Data Source: This registry will collect data from participants and healthcare providers involved in their care or the care of their infants via concise data collection forms at predefined timepoints during pregnancy, at pregnancy outcome, and up to 1 year of infant age.

Study Size: The registry aims to include as many pregnant individuals as possible, with no defined upper limit on enrollment in each cohort, to estimate the prevalence of the primary outcome, MCM, with meaningful confidence and precision. This approach aims to achieve adequate sample size to address additional research questions of interest, and/or maintain generalizability and representativeness of the registry population. Assuming a prevalence of MCM equivalent to 3% in each cohort, 1,143 and 303 live births in the analysis population of each cohort are needed to estimate the prevalence of MCM with ±1% and 2% precision, respectively.

Data Analysis: Participant characteristics will be summarized with descriptive statistics for each cohort. Comparative analyses will be conducted for each outcome if sample size permits. Supplementary analyses will be conducted that include pregnant individuals who were excluded from the analysis population. If sample size permits, subgroup and sensitivity analyses will be performed to examine the extent to which changes in certain methods or assumptions affect the results.

Milestones: The IBD-PR is expected to launch in March 2025, and the end of data collection is planned for 30 September 2032.

ELIGIBILITY:
Inclusion Criteria:

Exposed and unexposed cohort:

* A resident of the US or Canada at enrollment
* Currently pregnant
* 18 to 50 years of age at enrollment
* Physician-confirmed diagnosis of IBD (UC, CD, other and unspecified noninfective gastroenteritis and colitis [ICD-10 K52] and indeterminate colitis [ICD-10 K52.3])
* Evidence of a personally signed and dated informed consent document or, upon waiver of written consent by the relevant institutional review board (IRB)/independent ethics committee, verbal consent, indicating that the individual (or a legally acceptable representative) has been informed of all pertinent aspects of the study
* Authorize their HCP to provide data to the registry
* Provide contact information (for participant and HCPs)

Exposed cohort only:

- Exposed to an IBD pharmacotherapy during pregnancy

Exclusion Criteria:

Exposed and unexposed cohort:

* Exposure to methotrexate during pregnancy

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant individuals across the US & Canada who learn of the study via nationwide advertising campaigns or via their healthcare providers
Sampling Method: Non-Probability Sample
Enrollment: 832 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2032-09 (Estimated); Study Completion 2032-09 (Estimated)

PRIMARY OUTCOMES:
Major congenital malformation | Full pregnancy period (~9 months)
  An abnormality of body structure or function that is present at birth, is of prenatal origin (i.e., birth defect), has significant medical, social, or cosmetic consequences for the affected individual, and typically requires medical intervention.

SECONDARY OUTCOMES:
Minor congenital malformation | Full pregnancy period (~9 months)
  An anomaly or abnormality of body structure that is present at birth, is of prenatal origin (i.e., birth defect), poses no significant health problem in the neonatal period, and tends to have limited social or cosmetic consequences for the affected individual.
Spontaneous abortion | <20 gestational weeks
  An involuntary fetal loss or the expulsion of the products of conception occurring at <20 gestational weeks.
Pregnancy termination | Full pregnancy period (~9 months)
  A voluntary fetal loss or interruption of pregnancy that occurs for any reason, including but not limited to for the preservation of maternal health or because of fetal abnormalities.
Preeclampsia | Full pregnancy period (~9 months)
  A disorder of pregnancy associated with new-onset hypertension, which occurs most often after 20 weeks of gestation and frequently near term, and proteinuria. Or, in the absence of proteinuria, it is defined as new-onset hypertension with the new onset of any of the following:
  * Thrombocytopenia: platelet count <100,000/mL
  * Renal insufficiency: serum creatinine concentrations >1.1 mg/dL or a doubling of the serum creatinine concentration in the absence of other renal disease
  * Impaired liver function: elevated blood concentrations of liver transaminases to twice the normal concentration
  * Pulmonary edema
  * New-onset headache unresponsive to medication and not accounted for by alternative diagnoses or visual symptoms
Eclampsia | Full pregnancy period (~9 months)
  New-onset tonic-clonic, focal, or multifocal seizures in the absence of other causative conditions such as epilepsy, cerebral arterial ischemia and infarction, intracranial hemorrhage, or drug use.
Stillbirth | ≥20 gestational weeks
  Involuntary fetal loss occurring at ≥20 gestational weeks or, if gestational age is unknown, a fetus weighing ≥350g
Preterm birth | <37 gestational weeks
  A live birth occurring at <37 gestational weeks
Small for gestational age | At infant birth (up to 12 months of age)
  Birth weight <10th percentile for sex and gestational age using standard growth charts for full and preterm live-born infants.
Gestational diabetes | Full pregnancy period (~9 months)
  Any degree of glucose intolerance with onset or first recognition during pregnancy
Pregnancy induced hypertension | >20 gestational weeks
  A disorder of pregnancy defined as a systolic blood pressure of 140 mm Hg or more or a diastolic blood pressure of 90 mm Hg or more, or both, on two occasions at least 4 hours apart after 20 weeks of gestation in a woman with previously normal blood pressure
Placental abruption | Full pregnancy period (~9 months)
  Premature separation of the placenta from its uterine attachment before the delivery of a fetus
Postnatal growth deficiency | Up to 12 months of age
  Weight, length, or head circumference in <10th percentile for sex and chronological age using standard growth charts
Infant developmental delay | Up to 12 months of age
  Failure to achieve the developmental milestones for chronological age, as defined by the CDC.
Infant hospitalization | Up to 12 months of age
  The admission of an infant to a hospital
Infant infections (serious or nonserious) | Up to 12 months of age
  Infant infections that resulted in medical visit or hospitalization
Infant death | Up to 12 months of age
  The death of an infant before his or her first birthday

CONTACTS AND LOCATIONS:
Overall Officials: Ronna L Chan, PhD, MPH, Principal Investigator — PPD, Part of Thermo Fisher Scientific
Locations (1):
- PPD, Wilmington, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://ibdpregnancyregistry.com